CLINICAL TRIAL: NCT02688413
Title: Randomized Parallel-group Study Evaluating the Effectiveness and Cost-effectiveness of the Co-administration of MindMotionPRO Plus Standard Practice Versus Standard Practice in Early Post-stroke Upper-limb Rehabilitation
Brief Title: Study Evaluating the MindMotionPRO for Early Post-stroke Upper-limb Rehabilitation
Acronym: MOVE-Rehab
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: slow recruitment, evolution of investigational device, differences in healthcare models affecting trial
Sponsor: Mindmaze SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MindMaze-2016-RCT01
Record Dates: First submitted 2016-02-12; First posted 2016-02-23 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Stroke; Motor Disorders
Keywords: Virtual reality; Stroke; Neurorehabilitation; Upper-limb rehabilitation; Training games
MeSH Terms: conditions — Stroke; Motor Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MindMotionPRO (Experimental): MindMotionPRO exercises in addition to standard practice for upper limb rehabilitation
  Interventions: Device: MindMotionPRO
- Self-Directed Prescribed Exercises (Active Comparator): Self-Directed Prescribed Exercises in addition to standard practice for upper limb rehabilitation
  Interventions: Other: Self-Directed Prescribed Exercises

INTERVENTIONS:
Device: MindMotionPRO — The MindMotionPRO, a certified device for medical use, is a virtual reality based system to train upper limb activities in a game scenario. The participant will receive 5 exercises sessions with the MindMotionPRO per week over 4 weeks. This is done in addition to standard practice for upper limb rehabilitation which should be at least 30 min five times per week.
  Arms: MindMotionPRO
Other: Self-Directed Prescribed Exercises — GRASP is an arm and hand exercise program for stroke patients, designed to supplement standard rehabilitation therapies. The participant will receive 5 GRASP exercises sessions per week over 4 weeks. This is done in addition to standard practice for upper limb rehabilitation which should be at least 30 min five times per week.
  Other Names: Graded Repetitive Arm Supplementary Program (GRASP)
  Arms: Self-Directed Prescribed Exercises

SUMMARY:
Randomised controlled multi-centered study using MindMotionPRO, an immersive virtual reality based system for upper limb motor rehabilitation in early post-stroke patients. The study aims to evaluate the ability of MindMotionPRO technology to increase the rehabilitation dose. Effectiveness will be evaluated by validated rehabilitation performance scales. Cost-effectiveness will be assessed by the resource utilization.

DETAILED DESCRIPTION:
The goal of the study is to show that MindMotionPRO is a tool that allows a patient to increase the amount of rehabilitation therapy performed. This study will measure the rehabilitation dose, as measured by the duration of the rehabilitation session and the number of exercises performed by the patient. The study hypothesis is that patients in the MindMotionPRO group will spend more time performing rehabilitation exercises than in the Self-Directed Prescribed exercises group. The effectiveness of the MindMotionPRO versus Self-Directed Prescribed Exercises will also be measured, based on the change in rehabilitation performance measures. The cost-effectiveness will be measured by the resource utilization, as defined by the time spent by the therapist providing the rehabilitation session.

ELIGIBILITY:
Inclusion Criteria:

* Male/female > 18 years old
* First ever unilateral supratentorial ischemic stroke with contralateral upper extremity weakness
* 1 to 6 weeks post-stroke
* Able to give informed consent
* Not participating any other intervention studies
* Experiencing motor difficulties in using the paretic arm, with a FMA-UE score in the range of 20 to 40 out of 66
* Stroke severity with NIHSS score between 5 (mild) and 14 (moderate) out of 42
* The participant is expected to remain available (geographically stable) for 4 months after enrolment.

Exclusion Criteria:

* Any medical condition compromising the safety or the ability to take part to the study (such as insufficient vision or hearing, inability to participate to therapy session, inability to communicate, upper limb condition not linked to stroke, uncontrolled blood pressure, uncontrolled diabetes, co-morbidity)
* Recurrent and moderate to high upper limb pain limiting delivery of rehabilitation dose
* History of more than one epileptic seizures since stroke onset or uncontrolled epileptic seizure
* Mild to severe cognitive impairment (Mini mental state exam (MMSE) score < 24/30)
* Depression (Hospital Anxiety and Depression Scale > 8/21)
* Moderate to severe hemispatial neglect compromising the ability to take part to the study, as determined by the Bells tests (> 6 errors)
* Brain stem stroke

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Rehabilitation dose as measured by the duration of the rehabilitation session without planned rest periods | 4 weeks

SECONDARY OUTCOMES:
Number of exercises performed | 4 weeks
Change from Baseline in upper extremity motor function measured by the Fugl-Meyer Assessment for Upper Extremity (FMA-UE) and its subscales | baseline, 4 weeks, 16 weeks
Change from Baseline in upper extremity motor ability measured by the streamlined Wolf Motor Function Test (sWMFT) score | baseline, 4 weeks, 16 weeks
Change from Baseline in self-care ability measured by the Barthel index (BI) | baseline, 4 weeks, 16 weeks
Change from Baseline in functional independence measured by the Modified Ranking Scale (MRS) and associated disability-adjusted life year (DALY) | baseline, 4 weeks, 16 weeks
Change from Baseline in the general health status as measured by the Stroke Impact scale (SIS) | baseline, 4 weeks, 16 weeks
Change from Baseline in the severity of stroke symptoms as measured by the NIH stroke scale (NIHSS) | baseline, 4 weeks, 16 weeks
Change from Baseline in arm function in daily activities as measured by the Motor Activity Log (MAL) | baseline, 4 weeks, 16 weeks
Motivation measured by the Intrinsic Motivation Index (IMI) | 1 week and 4 weeks

OTHER OUTCOMES:
Resource utilization: time spent administrating rehabilitation exercises | 4 weeks
  therapist (physiotherapist or other medical staff) time spent administrating rehabilitation exercises
Change from Baseline in upper extremity muscle strength measured by the Medical research Council Scale (MRC) | Baseline, 1 week, 2 weeks, 3 weeks, 4 weeks and 16 weeks
  muscle strength for shoulder elevation, elbow flexion/extension, forearm pronation/supination and wrist extension/flexion

CONTACTS AND LOCATIONS:
Overall Officials: Valeria Caso, MD, Principal Investigator — Azienda Ospedale Santa Maria della Misericordia, Italy
Locations (3):
- Schön Klinik, Bad Aibling, Germany
- Santa Maria della Misericordia Hospital, Perugia, Umbria, Italy
- Queen Elisabeth University Hospital, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided